CLINICAL TRIAL: NCT00300170
Title: Determinants of Engagement in HIV Primary Care Services Among Black and Hispanic Single Room Occupancy Hotel Residents in New York City
Brief Title: Engagement in HIV Primary Care Services
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); CitiWide Harm Reduction (Other)
Responsible Party: Principal Investigator, Chinazo Cunningham, Prof Dept of Medicine, Montefiore Medical Center
Other Study IDs: 04-04-081
Record Dates: First submitted 2006-03-07; First posted 2006-03-08 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: HIV Infections; Unstable Housing
Keywords: HIV; race; unstable housing; health services accessibility; health services utilization; substance abuse; AIDS; health services research; social support; depression; trust; discrimination
MeSH Terms: conditions — HIV Infections; Patient Acceptance of Health Care; Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Depression

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study is to look at things that may affect whether or not people who are HIV-infected get into medical care and stay in medical care. some of the things that will be examined include how drug use, HIV disease severity, mental health, housing, trust, feelings of discrimination, social support, relationship with provider, and patient's race and provider's race are linked with whether or not people get health care. People who are enrolled in the study will be interviewed once, and their medical records will be examined.

DETAILED DESCRIPTION:
The purpose of this study is to understand the determinants of entry and engagement in HIV primary care services for Blacks and Hispanics living in single room occupancy (SRO) hotels in Bronx and Manhattan, NY. More specifically, the goal is to examine baseline cultural characteristics of the patient, health-related characteristics of the patient, the patient-provider relationship, and the impact of community outreach on engagement in health care. The objectives are to: examine the association between trust, relationship with provider, social support, and health beliefs with engagement in HIV primary care services; examine the association between health-related characteristics and engagement in HIV primary care services; examine the association of perceived cultural concordance between provider and patient with engagement in HIV primary care services; and, explore the relationship between community outreach and entry into HIV primary care services.

We will be recruiting a convenience sample of 500 Black or Hispanic HIV-infected adults living in 14 SRO hotels (transitional emergency housing) in the Bronx and Manhattan, NY. We will be conducting interviews through auditory computer-assisted self-interviewing (A-CASI) technology, using standardized research instruments administered in English or Spanish. We will also be reviewing medical charts and records from Citiwide and Montefiore appointment databases.

Understanding barriers to engagement in HIV primary care will lead to development of culturally relevant interventions to assist Black and Hispanic persons in entering and engaging in HIV treatment. Implementation of these interventions will ultimately help reduce disparities in HIV-related healthcare, as well as reduce HIV morbidity and mortality in Black and Hispanic populations.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age, HIV-infected, living in one of 15 different single room occupancy hotels in New York City, English or Spanish speaking

Exclusion Criteria:

* HIV-negative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2004-10; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Chinazo O Cunningham, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States